CLINICAL TRIAL: NCT02421653
Title: A Randomised Controlled Trial of Iodine-containing Micronutrient Powders Versus Oral Iodised Oil to Prevent Iodine Deficiency in Weaning Infants
Brief Title: RCT of Iodine-containing MNPs vs Oral Iodized Oil to Prevent Iodine Deficiency in Weaning Infants
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: UNICEF (Other); Global Alliance for Improved Nutrition (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: EK-2014-N-35; EK-2014-N-35 (Other: ETH Zuerich)
Record Dates: First submitted 2015-03-11; First posted 2015-04-21 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Iodine Deficiency Disorders
Keywords: Micronutrient powders; MNP; Weaning; Home fortification; Iodine; Iodine deficiency; Iodine Deficiency Disorder; IDD; Infant; Growth; Iodised oil
MeSH Terms: interventions — Iodized Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- MNP90 + INERT OIL (Experimental): Daily micronutrient powders (14 micronutrients) containing 90 µg iodine as potassium iodate plus one inert oil capsule without iodine at the study start;
  Interventions: Dietary Supplement: MNP90; Dietary Supplement: INERT OIL
- MNP45 + INERT OIL (Experimental): Daily micronutrient powders (14 micronutrients) containing 45 µg iodine as potassium iodate plus one inert oil capsule without iodine at the study start;
  Interventions: Dietary Supplement: MNP45; Dietary Supplement: INERT OIL
- IODISED OIL + INERT MNP (Experimental): Daily inert powder (maltodextrin, no micronutrients) plus one oral dose of 200 mg iodine as iodised poppy seed oil at the study start
  Interventions: Dietary Supplement: IODISED OIL; Dietary Supplement: INERT MNP
- NON-IODISED MNP + INERT OIL (Active Comparator): Daily micronutrient powders (14 micronutrients) without iodine plus one inert oil capsule without iodine at the study start.
  Interventions: Dietary Supplement: INERT OIL; Dietary Supplement: NON-IODISED MNP

INTERVENTIONS:
Dietary Supplement: MNP90 — 90 µg iodine-fortified micronutrient powder sachet (14 micronutrients); oral route; 1 daily
  Arms: MNP90 + INERT OIL
Dietary Supplement: MNP45 — 45 µg iodine-fortified micronutrient powder sachet (14 micronutrients); oral route; 1 daily
  Arms: MNP45 + INERT OIL
Dietary Supplement: IODISED OIL — 200 mg iodine oil capsule; oral route; once at study start
  Arms: IODISED OIL + INERT MNP
Dietary Supplement: INERT OIL — Non-iodised evening primrose oil capsule; oral route; once at study start
  Arms: MNP45 + INERT OIL; MNP90 + INERT OIL; NON-IODISED MNP + INERT OIL
Dietary Supplement: INERT MNP — Un-fortified powder sachet (maltodextrin, no micronutrients); oral route; 1 daily
  Arms: IODISED OIL + INERT MNP
Dietary Supplement: NON-IODISED MNP — Un-fortified micronutrient powder sachet (14 micronutrients); oral route; 1 daily
  Arms: NON-IODISED MNP + INERT OIL

SUMMARY:
In this study, two intervention strategies to address iodine deficiency and prevent iodine deficiency disorders in breast-fed weaning infants will be evaluated in a mild to moderate iodine-deficient population in Zamboanga del Norte, Philippines, Southeast Asia.

DETAILED DESCRIPTION:
Universal salt iodization (USI) is the most effective means to ensure optimal population iodine status and prevent iodine deficiency. In countries where USI is well implemented it is generally assumed that iodine requirements of infants are covered through breast milk. As infants wean from breast milk, at the age of 4-6 months, iodized salt programs likely contribute little to their iodine intakes. Home-prepared complementary foods have low native iodine content and pediatric guidelines recommend no extra salt be given to infants during the first year making the dietary sources of iodine limited. Weaning infants may therefore be particularly vulnerable to iodine deficiency and its effects.

Iodine is an essential micronutrient and an integral component of the thyroid hormones, needed for normal growth and development, particularly of the brain. Thyroid hormones play a critical role for development of the central nervous system from early fetal life until well after birth. Thyroid hormone insufficiency during postnatal development is associated with sensorimotor and language deficits and hypothyroidism in infancy is associated with poorer language, memory skills, fine motor, auditory processing, attention and executive processing.

In iodine deficient areas where iodized salt coverage is poor, WHO, UNICEF and the International Council for the Control of Iodine Deficiency Disorders (ICCIDD) recommend infants between 7 and 24 months be given a daily dose of 90 µg iodine (potassium iodate) or an annual dose of 200 mg iodine (iodised oil). The scientific evidence for this recommendation is weak, however, and it is uncertain under what conditions the two prevention strategies may be applied and which of the two is best when.

The objective of this study is to evaluate the efficacy and safety of the two recommended intervention strategies in iodine-deficient weaning infants. The need for high-quality controlled studies to better understand the potential contribution and synergy of alternative strategies to help achieve optimal iodine nutrition in different population groups and settings has recently been defined as a major research priority.

Following a cross-sectional, pilot study, we will conduct a randomized controlled trial to assess the efficacy of two daily doses of iodine as potassium iodate (90 µg, 100% of the WHO recommended dose, and 45 µg, 50% of the WHO recommended dose) and the annual dose of 200 mg iodine in iodised oil, via a randomized, controlled trial in weaning infants of lactating mothers living in an area affected by mild to moderate iodine deficiency in Zamboanga del Norte, Philippines, Southeast Asia.

We will compare the efficacy of each of the iodine doses against each other, and against micro-nutrients given alone, estimate the optimal level of iodine for inclusion in MNPs, and report on the safety of these interventions in weaning infants.

This study will provide important guidance to public health experts, governments and international organisations to ensure normal infant thyroid function and growth and development.

ELIGIBILITY:
Except for the infant age criteria, the selection and exclusion criteria are the same for all participants (pilot and intervention):

Inclusion criteria:

* Ages:
* For pilot - aged 6 - 18 months (+2 weeks, no infant < 6 months)
* For intervention - aged 6 - 9 months (+2 weeks, no infant < 6 months)
* Born to a healthy singleton pregnancy
* Term (week 38 to 42) delivery
* Family residence at the study site for at least 12 months prior to the start of the study and anticipated residence for at least a further 12 months (mother and infant)
* Exclusively breastfed for at least 2 months, or if not, having received no other sources of iodine intake (in formula, supplements, or foods)
* Signed informed consent

Exclusion criteria:

* Suffering from severe acute malnutrition(< 3 weight-for-height z-scores)
* Known history of medical illnesses
* Taking chronic medications (mother and infant)
* Use of iodine containing dietary supplements during the last 6 months (mother and infant)
* Exposure to iodine containing X-ray / CT contrast agent, skin disinfectants or medications during the last 6 months (mother and infant)
* Participation in any other clinical study (mother and infant) or participated in the pilot study (infant)

NB: Severe Acute Malnutrition is defined as being below 3 standard deviations (SD) of the WHO standard for weight-for-height ratio for infants and children aged 6 to 60 months. All infants identified with SAM will be excluded from the study and referred to hospital or nutrition clinic for treatment.

Ages: 6 Months to 9 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Infant urinary iodine concentration (UIC) | 24 weeks
Infant dried blood spot thyroglobulin (DBS-Tg) | 24 weeks

SECONDARY OUTCOMES:
Infant dried blood spot TSH (DBS-TSH) | 24 weeks
Infant dried blood spot total T4 (DBS-T4) | 24 weeks
Infant somatic growth (head circumference, weight, length) | 24 weeks, and if results significant at this point, 52 weeks
Thyroid autoimmunity | 24 weeks
  Measurement of thyroid antibodies
Safety (Composite measure of infant morbidities and infant mortality) | 24 weeks
  Composite measure of infant morbidities and infant mortality

OTHER OUTCOMES:
Infant urinary creatinine concentration | 24 weeks
Infant urinary sodium concentration | 24 weeks
Mother urinary iodine concentration (UIC) | 24 weeks
Mother breast milk iodine concentration (BMIC) | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Zimmermann, MD, Principal Investigator — ETH Zuerich